CLINICAL TRIAL: NCT01214213
Title: NON-SPECIFIC CHRONIC BACK PAIN; INSIGHT FROM SPATIAL ASPECTS OF LUMBAR SPINAL MUSCLE ACTIVATION
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Inge Ringheim, MSc, The Hospital of Vestfold
Other Study IDs: MULTI2009
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

SUMMARY:
There is evidence for altered muscle activity patterns in individuals with non-specific chronic back pain (NSCBP). It is unknown why these alterations in activation pattern occur and how they may be linked to pain experience and to the development of CNSBP. The main objective of this study is to investigate the spatial aspects of muscle activation in relation to fatigue/endurance and CNSBP. A novel approach, utilizing a new multi-channel surface-EMG (MCsEMG) technique will be applied in this project to get insight in fundamental mechanisms related to motor control and fatigue/endurance. In this project data from healthy persons and from patients with NSCBP will be collected and analyzed. NSCBP patients will be compared to healthy persons. To minimize heterogeneity between groups the subject's age range will be from 30 - 50 years. The investigators main hypothesis is that motor control mechanisms of the lumbar muscles are disturbed in NSCBP patients compared to normals, explaining the reduced tolerance for static postures. There has been little investigation of the lumbar musculature with MCsEMG recordings. The lumbar musculature has a complex organization; many, relatively small muscles, in a restricted area. Utilizing two HDsEMG grids with 252 Ag/AgCl contacts will be the superior non-invasive method to investigate motor control mechanisms in this region, and further the investigators understanding of neuromuscular adaptations related to NSCBP. The project may demonstrate changes that will lead us to new insight and new strategies for the treatment of back pain.

ELIGIBILITY:
Inclusion Criteria:

* patients
* diagnosed with chronic NSCBP >3 months duration
* healthy controls
* no back pain.

Exclusively exclusion criteria for this group will be back pain in the previous year or back pain lasting longer than one week in previous 3 years.

Exclusion Criteria:

* anamnesis of medical or drug abuse
* surgery on the musculoskeletal system of the trunk
* known congenital malformation of the spine or scoliosis
* body mass index >27 kg/m2
* systemic-neurological-degenerative disease
* history of stroke
* psychiatric disorder
* pregnancy and abnormal blood pressure.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Chronic non-spesific low back pain and healthy control subjects
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2009-09; Primary Completion 2014-01 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aage Indahl, Phd, Study Chair
Locations (1):
- Vestfold Hospital Trust, Kysthospitalet, Stavern, Norway